CLINICAL TRIAL: NCT00003109
Title: Phase I Pharmacokinetic and Pharmacodynamic Trial of Irinotecan in Combination With Tomudex in Patients With Refractory Solid Malignancies
Brief Title: Irinotecan Plus Raltitrexed in Treating Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065851; P30CA006927 (NIH); FCCC-96116 (Other: Fox Chase Cancer Center); NCI-T96-0113 (Other: National Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2004-07-08 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan; raltitrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: raltitrexed

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of irinotecan plus raltitrexed in treating patients who have refractory solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of irinotecan in combination with raltitrexed in patients with refractory solid tumors. II. Describe and quantify the toxic effects of this combination treatment regimen in a minimally pretreated patient population. III. Determine the pharmacokinetics of this combination treatment regimen. IV. Document any antitumor activity of this combination treatment regimen in this patient population.

OUTLINE: This is a dose escalation study of irinotecan and raltitrexed. Patients receive irinotecan IV over 90 minutes on days 1 and 8 followed by raltitrexed IV over 15 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients each receive escalating doses of irinotecan and raltitrexed until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Additional cohorts receive raltitrexed on day 2 rather than day 1 near the final dose levels of the combination drugs.

PROJECTED ACCRUAL: A maximum of 36 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven malignant solid tumor that has failed prior conventional chemotherapy or for which no established therapy exists Recurrent or metastatic gastrointestinal adenocarcinoma with no prior therapy eligible No evidence of CNS metastases (brain or leptomeningeal disease)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,500/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.8 mg/dL SGOT and SGPT less than 3 times upper limit of normal (ULN) Alkaline phosphatase less than 3 times ULN (5 times ULN for metastatic disease) Renal: Creatinine no greater than 1.8 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No congestive heart failure Other: No uncontrolled diabetes Not pregnant or nursing Negative pregnancy test No other serious medical illness (e.g. clinically active infectious process) No psychiatric illness precluding study No ascites or pleural effusion

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No more than 1 prior adjuvant chemotherapy regimen No more than 1 prior chemotherapy regimen for recurrent or metastatic disease No prior irinotecan or raltitrexed At least 8 weeks since prior nitrosourea or mitomycin and recovered Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Prior radiotherapy limited to no greater than 25% of bone marrow Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1997-12; Primary Completion 2000-10 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal J. Meropol, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States